CLINICAL TRIAL: NCT03959553
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Design, Prospective, Phase IIa Clinical Trial to Evaluate the Safety and Efficacy of GV1001 Administered Subcutaneously for the Treatment of Moderate Alzheimer's Disease
Brief Title: GV1001 Subcutaneous(SC) for the Treatment of Moderate Alzheimer's Disease (AD)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped due to protocol amendment and project name change.
Sponsor: GemVax & Kael (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KG7/2017
Record Dates: First submitted 2019-05-08; First posted 2019-05-22 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2019-05

CONDITIONS: Moderate Alzheimer's Disease
Keywords: Alzheimer's Disease; GV1001
MeSH Terms: conditions — Alzheimer Disease | interventions — GV1001 peptide; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo SC injection administered once weekly for 4 weeks then every 2 weeks through Week 24
  Interventions: Drug: Normal saline
- GV1001 0.56 mg (Experimental): GV1001 0.56 mg SC injection administered once weekly for 4 weeks then every 2 weeks through Week 24
  Interventions: Drug: GV1001
- GV1001 1.12 mg (Experimental): GV1001 1.12 mg SC injection administered once weekly for 4 weeks then every 2 weeks through Week 24
  Interventions: Drug: GV1001

INTERVENTIONS:
Drug: GV1001 — Lyophilized peptide from hTERT
  Other Names: Tertomotide
  Arms: GV1001 0.56 mg; GV1001 1.12 mg
Drug: Normal saline — 0.9% normal saline
  Arms: Placebo

SUMMARY:
The current study is being conducted by the Sponsor to evaluate the efficacy and safety of GV1001 (0.56 mg and 1.12 mg) administered subcutaneously as a treatment for moderate Alzheimer's disease (AD). GV1001 has been shown to inhibit neurotoxicity, apoptosis, and the production of reactive oxygen species induced by amyloid beta in neural stem cells by mimicking the extra-telomeric functions of human telomerase reverse transcriptase (hTERT). In nonclinical studies, using both mild (early stage) and severe (late stage) AD mouse models, GV1001 has been shown to improve cognitive function and memory, as well as significantly reduce the amount of amyloid beta and tau proteins. The multifunctional effect of GV1001 makes it a promising therapeutic option for the treatment for AD.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, dose finding, parallel-group Phase IIa study in participants with moderate AD. The study population will be comprised of male and female participants between 55 and 85 years of age, inclusive, with a diagnosis of probable AD based on National Institute of Neurological and Communicative Disorders and Stroke-Alzheimer's Disease and Related Disorders Association (NINCDS ADRDA) criteria. Participants must also meet Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria for dementia and have an Mini-Mental State Examination (MMSE) score ≥10 to <20. Participants or their legal representative, as well as the participant's caregiver, must be able to provide written informed consent.

The study will consist of a screening visit (up to 4 weeks prior to first dose), a 26-week double blind treatment period, and an end-of-study (EOS) visit. In the event a participant discontinues treatment or the study prematurely, the participant will be asked to return for an early termination (ET) visit for safety assessments. These assessments are the same as those done at the EOS visit.

Prior to randomization, eligibility of potential participants will be confirmed through an adjudication process in which screening data (eg, MMSE) obtained to evaluate AD status are reviewed by a central independent adjudicator. The adjudicator will review the scoring sheet completed by the Investigator prior to randomization and provide an independent assessment of the participant's eligibility and may request exclusion of a participant from entry into the study. A central independent reader will review magnetic resonance imaging (MRI) or computed tomography (CT) scans or reports to confirm eligibility. Investigators must not randomize a participant prior to receipt of this independent confirmation of the participant's eligibility.

Eligible participants will be randomized to treatment with either GV1001 0.56 mg, GV1001 1.12 mg, or placebo (normal saline) in a 1:1:1 ratio. Study treatment (GV1001 0.56 mg, GV1001 1.12 mg, or placebo) will be administered by subcutaneous (SC) injection every week for 4 weeks (4 times) followed by SC administration every 2 weeks through Week 24 (10 times) for a total of 14 SC administrations of study treatment.

Efficacy evaluations will be performed at baseline, Week 12, and Week 26 using the Mini-Mental State Examination (MMSE), Alzheimer's Disease Assessment Scale-cognitive (ADAS cog), Clinician's Interview-Based Impression of Change (CIBIC)-Plus, Clinical Dementia Rating - Sum of Boxes (CDR-SB), Alzheimer's Disease Cooperative Study-Activities of Daily Living scale (ADCS-ADL), and Neuropsychiatric Inventory (NPI) scales. The efficacy evaluations are to be done in the same order at each visit. To ensure the objectivity and accuracy of the study results, efficacy evaluations must be performed by adequately trained and experienced clinicians. The raters must be certified for this study to administer the Mini-Mental State Examination (MMSE), Alzheimer's Disease Assessment Scale-cognitive (ADAS cog), Clinician's Interview-Based Impression of Change (CIBIC)-Plus, Clinical Dementia Rating - Sum of Boxes (CDR-SB), Alzheimer's Disease Cooperative Study-Activities of Daily Living scale (ADCS-ADL), and Neuropsychiatric Inventory (NPI) scales. Training, certification, and materials for rating will be provided by a rater training group. To mitigate the risk of breaking the blind, the efficacy evaluator is not to be involved in the participant's treatment or have access to the record of reported Adverse Events (AEs).

Safety will be assessed throughout the study by monitoring for AEs, laboratory evaluations, electrocardiogram (ECG) findings, vital sign measurements, and suicidal ideation and behavior (C-SSRS). Pharmacodynamics will be evaluated by collecting blood and cerebrospinal fluid (CSF) for analysis of biomarkers of AD. Blood samples will also be collected for pharmacokinetic (PK) and immunogenicity analysis, including determination of GV1001 plasma concentrations (sparse PK) and antibodies to GV1001.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 55 to 85 years of age, inclusive, at the time of signing the informed consent.
2. Diagnosis of probable AD based on NINCDS-ADRDA criteria.
3. Diagnosis of dementia based on DSM-V criteria.
4. Moderate dementia as evidenced by MMSE score ≥10 to <20 at screening.
5. Magnetic resonance imaging or CT within 12 months prior to randomization with findings consistent with AD and without any other disease that may cause dementia.
6. If receiving an FDA-approved medication for AD (ie, donepezil, galantamine, rivastigmine, memantine, or memantine/donepezil combination product) must be on a stable dose for at least 3 months prior to screening visit.
7. If receiving an OTC supplement for cognition (eg, gingko biloba, omega-3 polyunsaturated fatty acid, vitamin E, curcumin) must be taking a stable dose for at least 3 months prior to screening visit.
8. Able to visit the study center and undergo cognitive, functional, and other tests specified in the protocol.
9. Has a caregiver who:

   * Agrees to accompany the participant to all study visits and able to supervise the participant's compliance with the study procedures and provide detailed information about the participant.
   * Either lives with the participant or sees the participant on average for ≥1 hours/day ≥3 days/week, or in the Investigator's opinion, the extent of contact is sufficient to provide meaningful assessment of changes in participant behavior and function over time and provide information on safety and tolerability.
   * Is able to read, understand, and speak the designated language at the study center.
   * Caregiver must be cognitively able to fulfill the requirements of the study.
10. A male participant must agree to use a highly effective contraception as detailed in Appendix 4 of this protocol during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period.
11. A female participant is eligible to participate if she is not pregnant (see Appendix 4), not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) as defined in Appendix 4. OR
    * A WOCBP who agrees to follow the contraceptive guidance in Appendix 4 during the treatment period and for at least 3 months after the last dose of study treatment.
12. A WOCBP must have a negative serum pregnancy test (beta human chorionic gonadotropin [β-hCG]) at screening and a negative urine pregnancy test at Visit 2 before randomization.
13. Written informed consent provided by participant or legal representative and caregiver prior to any study-specific procedures.

Exclusion Criteria:

1. Any other cause of dementia shown by MRI/CT findings and neurological examination within 12 months of randomization.

   * Possible, probable, or definite vascular dementia according to the National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherché et l'Enseignement en Neurosciences (NINDS-AIREN) criteria.
   * Evidence of significant abnormality that would suggest another potential etiology for dementia (eg, evidence of cerebral contusion, encephalomalacia, aneurysm, vascular malformation, >5 microhemorrhages, macrohemorrhage, single infarct >1cm3).
   * Other central nervous system diseases that may cause cognitive impairment (eg, cerebrovascular disease including cerebrovascular dementia, Parkinsonism, Huntington's disease, subdural hematoma, normal pressure hydrocephalus, brain tumor, Creutzfeldt-Jakob disease).
2. Concurrent or history of clinically significant psychiatric conditions (eg. Schizophrenia or bipolar affective disorder) that in the Investigator's opinion prevents the participant from participating, or is likely to confound interpretation of drug effect or affect cognitive assessments.
3. Vitamin B12, folic acid, syphilis serology, and thyroid stimulating hormone (TSH) results that are thought to contribute to the severity of dementia or cause dementia. Participants may be enrolled if in the Investigator's medical judgment the abnormal laboratory values are not the cause of the cognitive symptoms.
4. History of known or suspected seizures including febrile seizures (excluding self-limited childhood febrile seizures), a history of significant head trauma with loss of consciousness or recent unconsciousness that is not explained.
5. Acute or unstable cardiovascular disease, active peptic ulcer, uncontrolled hypertension, uncontrolled diabetes or insulin dependent patients or any medical condition that may interfere with the completion of the clinical study.
6. Known allergies, hypersensitivity, or intolerance to GV1001 or similar products or excipients.
7. History of alcohol, substance abuse or dependence as per DSM-V criteria (except nicotine dependence) within the last 2 years.
8. Concurrent malignancies or invasive cancers diagnosed within the past 5 years except for non-metastatic basal cell carcinoma or squamous cell carcinoma of skin, in situ carcinoma of the uterine cervix or non-metastatic prostate cancer
9. Sexually-active WOCBP or man capable of fathering a child who do not consent to using medicinally acceptable contraception (such as surgical sterilization, intrauterine contraceptive device, condom or diaphragm, an injectable or inserted contraceptive) during the study and for 3 months after the last dose of study treatment.
10. Pregnant, breast feeding, or planning a pregnancy or fathering a child while enrolled in the study or for 3 months after the las dose of study treatment.
11. Use of anxiolytics, narcotics, or sleep aids in a manner that would interfere with cognitive testing, in the opinion of the Investigator. Atypical antipsychotics may be used at the discretion of the Investigator. Tricyclic antidepressants and monoamine oxidase (MAO) inhibitors are prohibited.
12. Previous treatment with GV1001.
13. Received an investigational product for AD within last 6 months.
14. Participated in another clinical study within 4 weeks prior to this study.
15. Renal impairment (creatinine clearance [CrCL] <30 mL/min).
16. Severe liver dysfunction (alanine aminotransferase [ALT] or aspartate aminotransferase [AST] >2 times the upper limit of normal [ULN]).
17. Body weight ≤35 kg.
18. Resides in a moderate to high dependency continuous care facility (residence in low grade assisted living facility where there is sufficient autonomy to permit valid evaluation of activities of daily living is allowed).
19. Any other reason that in the opinion of the Investigator would make the participant ineligible to participate or to complete this study.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognitive (ADAS-cog) | Week 26
  The proportion of participants with any improvement in ADAS-cog compared to the baseline and Week 26

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognitive (ADAS cog) | Week 26
  Change from baseline in ADAS cog at Week 26
Clinician's Interview-Based Impression of Change (CIBIC)-Plus | Week 26
  Change from baseline in CIBIC-Plus at Week 26
Clinical Dementia Rating - Sum of Boxes (CDR-SB) | Week 26
  Change from baseline in CDR-SB at Week 26
Alzheimer's Disease Cooperative Study-Activities of Daily Living (ADCS-ADL) | Week 26
  Change from baseline in ADCS-ADL at Week 26
Neuropsychiatric Inventory (NPI) | Week 26
  Change from baseline in NPI at Week 26
Mini-Mental State Examination (MMSE) | Week 26
  Change from baseline in MMSE at Week 26

IPD SHARING:
Plan to Share IPD: No